CLINICAL TRIAL: NCT04752878
Title: The Turkish Version Of The Ottawa Sitting Scale: Its Cultural Adaptation, Validation And Reliability In Patients Wıth Stroke
Brief Title: Turkish Version of Ottawa Sitting Scale in Patients With Stroke
Status: Completed | Type: Observational
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Mustafa Ertuğrul Yaşa, Assistant professor, Gulhane School of Medicine
Other Study IDs: 2020-363
Record Dates: First submitted 2021-02-05; First posted 2021-02-12 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Fall Due to Loss of Equilibrium; Acute Stroke; Balance; Distorted; Fear
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ottawa sitting scale — The Ottawa Sitting Scale is a performance-based balance measurement consisting of 10 items that aims to evaluate the sitting balance in a comprehensive, specific, efficient and functional manner.

SUMMARY:
The aim of the study is to describe the cultural adaptation of the Ottawa Sitting Scale and to examine the factor structure, reliability and validity of the scale in patients with stroke.

The scale will be translated into Turkish language by following the procedure. 80 patients will be recruited in the study. Berg Balance Scale and Trunk Impairment Scale will be included with Turkish Ottawa Sitting Scale to test the validity. Outcome measures will be repeated by a second physiotherapist the day after the first assessment for interrater reliability and conducted twice within 2 weeks (test-retest) for reliability.

The interrater and intrarater reliability of the Ottawa sitting scale will be determined using intraclass correlation coefficients and internal consistency will be assessed using Cronbach's alpha.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with acute stroke
* aged above 18 years

Exclusion Criteria:

* Patients who do not cooperate enough to read or approve the consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age diagnosed with acute ischemic or hemorrhagic stroke
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Ottawa sitting scale | Measurements will start with the first patient hospitalized (estimated in March 2021) and end with the evaluation of the 80th patient (estimated period of 12 months)
  A balance measurement scale for acute stroke patients. The scale tests the patient on a total of 10 items while sitting, with 5 items with eyes open and 5 items with eyes closed. An ordered scale (0-4) is used to score each item. The total score range of the scale is 0-40. Higher scores indicate a better outcome

SECONDARY OUTCOMES:
Berg balance scale | Measurements will start with the first patient hospitalized (estimated in March 2021) and end with the evaluation of the 80th patient (estimated period of 12 months)
  A balance measurement to determine the risk of falls. The scale consists of 14 items. Each item is scored between 0 and 4. 4 points indicate the ability to complete the task independently, 0 points indicate the failure to start the task. According to the scores, the cases are divided into groups as "high risk of falling (0-20 points)", "moderate fall risk (21-40 points)", "low risk of falling (41-56 points)" and the highest score 56 is considered to show the best balance
Trunk Impairment scale | Measurements will start with the first patient hospitalized (estimated in March 2021) and end with the evaluation of the 80th patient (estimated period of 12 months)
  A scale to evaluate motor disorders in the trunk after stroke. This scale consists of 3 sub-sections and 17 items that evaluate static sitting balance, dynamic sitting balance and coordination. The maximum score of the test is 40 points. High scores indicate good balance

CONTACTS AND LOCATIONS:
Locations (1):
- Sağlık Bilimleri Üniversitesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No